CLINICAL TRIAL: NCT03973294
Title: Assessment of Regional Lung Ventilation Distribution During Supraglottic and Subglottic Jet Ventilation by Electrical Impedance Tomography (EIT).
Brief Title: Assessment of Regional Lung Ventilation Distribution During Supraglottic and Subglottic Jet Ventilation by EIT.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Marita Windpassinger M.D., Principal Investigator, Medical University of Vienna
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 1298/2019
Record Dates: First submitted 2019-06-01; First posted 2019-06-04 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Respiratory Physiological Phenomena
Keywords: jet ventilation; electroimpedance tomography; supraglottic jet ventilation; subglottic jet ventilation

STUDY DESIGN:
Intervention Model Description: Patients undergoing elective micro laryngeal surgery will be assigned to subglottic JV via the new LaserJet catheter and supraglottic JV via the jet laryngoscope vice versa. The sequence of JV modes will be randomized (subglottic followed by supraglottic or supraglottic followed by subglottic JV).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supraglottic jet ventilation (Active Comparator): Ventilation of the patient is performed over a steel laryngoscope or a thin catheter by means of jet ventilation (JV) using the TwinStream jet ventilator (C. Reiner Corp, Vienna, Austria). The driving pressure of the device is 1.5-3 bar and respiratory rates of 10-900 per min can be provided. In superimposed high frequency jet ventilation (SHFJV), jet ventilation of normal frequency and high frequency is conducted simultaneously and enables ventilation at two different pressure levels through the steel jet laryngoscope. It is equipped with two jet nozzles, which are placed at the distal end of the jet laryngoscope.
  Interventions: Device: EIT-measurement
- Subglottic jet ventilation (Active Comparator): Subglottic HFJV is performed through the LaserJet catheter. It is characterized by the delivery of small tidal volumes from a high pressure jet at very high frequencies (100-400) followed by passive expiration for a very short period before delivering the next jet, creating an "auto-PEEP".
  Interventions: Device: EIT-measurement

INTERVENTIONS:
Device: EIT-measurement — The use of electrical impedance tomography (EIT) (SentecTom BB2, Landquart, Switzerland) allows the investigators to obtain a visual and quantitative representation of the areas of ventilation and aeration of the lung. The fundamental principle of lung EIT relies on the application of small alternating electrical currents into the thorax and voltage measurements using electrodes on the skin surface generating cross-sectional images representing impedance change in a slice of the thorax. It is a radiation-free imaging method which has the advantage to reveal real-time information.
  An array of electrodes (textile belt with 32 integrated electrocardiographic electrodes) has to be placed around the thorax to inject currents and to measure the resulting voltages on the thoracic surface.

SUMMARY:
Objective: To estimate regional lung volume changes by electrical impedance tomography (EIT) during supra- and subglottic jet ventilation via the jet laryngoscope and LaserJet catheter for performing laryngotracheal surgery.

Design: A monocentric, prospective, randomized study. Patients: Patients who require elective micro laryngo-tracheal surgery under jet ventilation.

Interventions: Patients undergoing elective micro laryngeal surgery will be assigned to subglottic JV via the new LaserJet catheter and supraglottic JV via the jet laryngoscope vice versa. The sequence of JV modes will be randomized (subglottic followed by supraglottic or supraglottic followed by subglottic JV). Hemodynamic and ventilation parameters will be monitored. Arterial blood gas samples will be drawn and the regional ventilation distribution assessed, using the EIT.

Outcomes measures: Reported EIT data of regional ventilation distribution, values of oxygenation and carbon dioxide elimination during the application of supra- and subglottic JV via jet laryngoscope and LaserJet catheter in patients undergoing laryngo-tracheal surgery. The purpose of this study is to investigate the influence of supraglottic and subglottic JV compared to standardized, controlled mask ventilation on measurements of pulmonary regional ventilation distribution by EIT, blood gas analyses and serological biomarkers.

DETAILED DESCRIPTION:
Surgical procedures of the larynx and trachea present special challenges for surgeons and anesthesiologists. To enable an unrestricted view of the operating field, ventilation of the patient is not performed over an endotracheal tube but instead over a steel laryngoscope or a thin catheter with Jet ventilation (JV). This enables precision surgical work, good visibility of the operating area and the safe use of various laser types. Over the last decades, different modalities of JV for laryngo-tracheal surgery have been developed. The former techniques of the supraglottic approach were improved with simultaneously applied low-frequency jet ventilation additionally to the high-frequency jet ventilation, called superimposed high-frequency jet ventilation (SHFJV). The SHFJV was developed in 1990 and was applied in several clinical trials [1-4] In recent years, a number of new catheters have been developed for the trans laryngeal subglottic approach of JV, like the translaryngeal Hunsaker MonJet Ventilation catheter and its successor, the LaserJet catheter. These catheters though can be used only with the HFJV. They provide less vocal cord movement and precise surgical manipulation are possible on one side, but on the other the risk of barotrauma may result in cases of proximal obstruction of the catheter.

[5, 6] Although jet ventilation is an established method to replace patients breathing during otorhinolaryngeal surgery, research is still required on efficient lung protective ventilation in order to provide adequate carbon dioxide (CO2) elimination, adequate oxygenation and in preventing ventilator induced lung injury. Jet ventilation techniques and access routes The TwinStream jet ventilator (C. Reiner Corp, Vienna, Austria) is routinely used for high-frequency jet ventilation (HFJV) or SHFJV in case of tubeless jet laryngoscopy (laryngeal micro- and laser surgery) and tracheoscopy. The device consists of two simultaneously operating ventilation units which can be adjusted separately. The driving pressure of the device is 1.5-3 bar and respiratory rates of 10-900 per min can be provided. Supraglottic jet laryngoscope In SHFJV, jet ventilation of normal frequency and high frequency is conducted simultaneously and enables ventilation at two different pressure levels through the steel jet laryngoscope. It is equipped with two jet nozzles, which are placed at the distal end of the jet laryngoscope, with the low-frequency jet stream passing the distal cannula, and the high-frequency jet stream at the proximal cannula. A third cannula at the tip of the laryngoscope allows ventilation pressure monitoring. The jet laryngoscope is introduced by the surgeon, for examining and operating structures within the laryngotracheal system. Supraglottic JV causes more laryngeal movement induced by disturbances through the high frequent inspiratory air passing the operating field compared to the subglottic jet ventilation. [9] Furthermore it leads to greater dryness of the vocal cords. During supraglottic SHFJV the escaping exhaled gases vent blood and secretion outward, reducing the risk of fluid aspiration and of displacing cells of any entity down to the tracheobronchial tree.

Advantages of SHFJV with the supraglottic inserted steel laryngoscope:

* Unlimited surgical access and vision of the operating field
* Laser resistant
* Protection of the airway through the inherent 'auto-PEEP (positive endexpiratory pressure)' effect
* Prevention of CO2 retention, lung alveolar collapse and improvement of the oxygen index Subglottic LaserJet Catheter Through the LaserJet catheter ventilation is performed only with HFJV. It is characterized by the delivery of small tidal volumes from a high pressure jet at very high frequencies (100-400) followed by passive expiration for a very short period before delivering the next jet, creating an "auto-PEEP".

The LaserJet catheter (C. Reiner Corp, Vienna, Austria) is made of polyterafluoroethylene and is non inflammable and provides a good micro anatomical overview of the operating structures [7,8,9] However, the LaserJet catheter is not laser resistant in regards of deformation damage (perforation) under direct exposure to a continuous laser beam. The use of the new 445 nm wavelength laser, the 'blue laser' eases the surgical performance by securing important laryngeal functionality even in advanced disease [3,4,10] While the exposure of the complete pathology is visualized and treated, the surrounding tissue is not dislocated or deformed.

[11] The LaserJet catheter has the advantage of minimizing movements of the larynx and vocal cords and facilitates the precise use of the blue laser without affecting healthy tissue.

Electrical impedance tomography (EIT) When evaluating different JV devices and techniques, tidal volume and minute ventilation are difficult to assess because SHFJV and HFJV are applied in an open airway system. Air entrainment occurs to a varying extent depending on the route of JV administration, anatomical factors and jet alignment with the airway. [13] A standard intraoperative monitoring does not provide accurate predictions about changes in regional lung ventilation. The use of electrical impedance tomography (EIT) (SentecTom BB2, Landquart, Switzerland) allows the investigators to obtain a visual and quantitative representation of the areas of ventilation and aeration of the lung. The fundamental principle of lung EIT relies on the application of small alternating electrical currents into the thorax and voltage measurements using electrodes on the skin surface generating cross-sectional images representing impedance change in a slice of the thorax. It is a radiation-free imaging method which has the advantage to reveal real-time information.

An array of electrodes (textile belt with 32 integrated electrocardiographic electrodes) has to be placed around the thorax to inject currents and to measure the resulting voltages on the thoracic surface. Analyzing EIT measurements during ongoing mechanical JV is a useful tool to detect imbalances in regional lung ventilation and in further consequence enables to optimize ventilator setting during surgery. The investigators will assess changes in regional lung ventilation distribution during supra- and subglottic JV compared to controlled mask ventilation. EIT, as a non-invasive method, may become a useful tool for adjustment of optimal positioning of the JV devices and for decision-making of the optimal type of the JV device (supraglottic laryngoscope versus subglottic jet catheter) by detecting atelectasis as "silent spaces" or over distension. This additional source of information could help fine tune the jet ventilator. Its intraoperative use could provide the basis for individual optimization of jet ventilator settings, especially in patients at risk for ventilation-perfusion mismatch and impaired gas exchange. Serological biomarkers of lung damage and inflammation It is still an open question whether the type of specific mechanical ventilation like HFJV and SHFJV have an influence on changes in serological biomarkers for lung damage and inflammation like Surfactant proteins (SP)-D [14-16], Krebs van den Lungen (KL)-6 [17, 18], Clara cell protein (CC16) [19, 20], Adrenomedullin (ADM) [21] or Interleukin 6 (IL-6) and 8 (IL-8). Studies revealed that in patients with normal lungs, relatively short periods of mechanical ventilation induce lung inflammation and that these changes depend on the ventilatory parameters applied. [22-25] The investigators will study the influence of JV on these serum levels in patients undergoing elective laryngotracheal surgery. Specific aims and hypotheses The objective of this study is to compare regional ventilation distribution, blood gas oxygenation, CO2 elimination and serum biomarkers with different jet ventilatory techniques and access routes.

Our primary aim is to determine whether supraglottic JV with the jet laryngoscope leads to a shift of the Center of Ventilation (COV) towards the ventral lungs compared to mask ventilation.

The secondary objective of the study is to investigate changes in ventro-dorsal ventilation distribution, measured as ventro-dorsal COV shift, under subglottic JV compared to standardized, controlled mask ventilation. Further study objectives are the comparison of ventilation distribution parameters between the two JV techniques, supra- and subglottic JV, and the analysis of oxygenation and CO2 elimination during these two ventilation modes over time. Furthermore, special serum biomarkers of pulmonary lung damage are determined after JV application. Primary hypothesis The primary hypothesis is that during the use of supraglottic jet ventilation, the COV is shifted to more ventrally located (non-dependent) lung sections compared to controlled mask ventilation.

Secondary hypothesis The secondary hypothesis is that subglottic JV ventilation leads to a ventral displacement of the COV compared to controlled mask ventilation and that this occurs to a greater extent than during supraglottic JV. Null hypothesis There is no significant displacement of COV into ventrally located lung sections under supraglottic jet ventilation compared to controlled mask ventilation.

ELIGIBILITY:
Inclusion Criteria

* Patients undergoing elective micro-laryngotracheal surgery
* Ventilation type: SHFJV and HFJV
* Jet devices: Jet laryngoscope and LaserJet catheter
* ASA 1-3
* Age 18- 99 years.

Exclusion Criteria

* acute bleeding in the area of the larynx/trachea
* infectious lung disease (e.g. tuberculosis)
* inability to perform retroflexion of the head (laryngoscope cannot be positioned properly)
* thoracic wall deformities
* obesity, BMI >30kg/m2
* implantable electronic devices (f.e. pacemaker, ICD)
* emergency surgery
* expected postoperative mechanical ventilation (Intensive Care Unit)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-06-07 (Actual); Primary Completion 2023-08-21 (Actual); Study Completion 2023-08-21 (Actual)

PRIMARY OUTCOMES:
Center of ventilation (COV) | The EIT measurements will be recorded on arrival in the operating room (OR) under spontaneous breathing, during standardized, controlled mask ventilation and 5 minutes after supra- and subglottic JV.
  Our primary aim is to determine whether supraglottic JV with the jet laryngoscope leads to a shift of the Center of Ventilation (COV) towards the ventral lungs compared to mask ventilation.

SECONDARY OUTCOMES:
ROI 1-4 | The EIT measurements will be recorded on arrival in the operating room (OR) under spontaneous breathing, during standardized, controlled mask ventilation and 5 minutes after supra- and subglottic JV.
  Sum of impedance changes in predefined regions of interest (ROI) 1-4
ΔEELI | The EIT measurements will be recorded on arrival in the operating room (OR) under spontaneous breathing, during standardized, controlled mask ventilation and 5 minutes after supra- and subglottic JV.
  Changes in end expiratory lung impedance
silent spaces | The EIT measurements will be recorded on arrival in the operating room (OR) under spontaneous breathing, during standardized, controlled mask ventilation and 5 minutes after supra- and subglottic JV.
  Areas with impedance changes <10%.
Blood gas analysis values | Blood will be drawn during mask ventilation, 5 minutes after supraglottic and 5 minutes after subglottic JV and at the end of surgery, before leaving to the recovery room for gas analysis and serum biomarkers.
  PaO2 (mmHg), PaCO2 (mmHg), PaO2/FiO2 index) are investigated over time during mask ventilation, supra- and subglottic JV
Special serum biomarkers for pulmonary inflammation and parenchyma damage | Blood will be drawn during mask ventilation, 5 minutes after supraglottic and 5 minutes after subglottic JV and at the end of surgery, before leaving to the recovery room for gas analysis and serum biomarkers.
  IL-6, IL-8, SP-D, KL-6, CC16, ADM) are determined preoperatively and postoperatively at fixed points

CONTACTS AND LOCATIONS:
Overall Officials: Marita Windpassinger, MD, MBA, Principal Investigator — Medical University of Vienna; Olga Plattner, MD, Study Director — Medical University of Vienna
Locations (1):
- Medical University Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bacher A, Lang T, Weber J, Aloy A. Respiratory efficacy of subglottic low-frequency, subglottic combined-frequency, and supraglottic combined-frequency jet ventilation during microlaryngeal surgery. Anesth Analg. 2000 Dec;91(6):1506-12. doi: 10.1097/00000539-200012000-00039. PMID 11094009
- [Background] Bacher A, Pichler K, Aloy A. Supraglottic combined frequency jet ventilation versus subglottic monofrequent jet ventilation in patients undergoing microlaryngeal surgery. Anesth Analg. 2000 Feb;90(2):460-5. doi: 10.1097/00000539-200002000-00041. PMID 10648340
- [Background] Lanzenberger-Schragl E, Donner A, Grasl MC, Zimpfer M, Aloy A. Superimposed high-frequency jet ventilation for laryngeal and tracheal surgery. Arch Otolaryngol Head Neck Surg. 2000 Jan;126(1):40-4. doi: 10.1001/archotol.126.1.40. PMID 10628709
- [Background] Rezaie-Majd A, Bigenzahn W, Denk DM, Burian M, Kornfehl J, Grasl MCh, Ihra G, Aloy A. Superimposed high-frequency jet ventilation (SHFJV) for endoscopic laryngotracheal surgery in more than 1500 patients. Br J Anaesth. 2006 May;96(5):650-9. doi: 10.1093/bja/ael074. Epub 2006 Mar 30. PMID 16574723
- [Background] Davies JM, Hillel AD, Maronian NC, Posner KL. The Hunsaker Mon-Jet tube with jet ventilation is effective for microlaryngeal surgery. Can J Anaesth. 2009 Apr;56(4):284-90. doi: 10.1007/s12630-009-9057-2. Epub 2009 Feb 25. PMID 19296189
- [Background] Frochaux D, Rajan GP, Biro P. [Laser-resistance of a new jet ventilation catheter (LaserJet) under simulated clinical conditions]. Anaesthesist. 2004 Sep;53(9):820-5. doi: 10.1007/s00101-004-0717-x. German. PMID 15448938
- [Background] Friedrich G, Mausser G, Gugatschka M. [Jet ventilation in laryngotracheal surgery]. HNO. 2008 Dec;56(12):1197-206. doi: 10.1007/s00106-008-1725-y. German. PMID 19020846
- [Background] Wegrzynowicz ES, Jensen NF, Pearson KS, Wachtel RE, Scamman FL. Airway fire during jet ventilation for laser excision of vocal cord papillomata. Anesthesiology. 1992 Mar;76(3):468-9. doi: 10.1097/00000542-199203000-00022. No abstract available. PMID 1539860
- [Background] Rubin JS, Patel A, Lennox P. Subglottic jet ventilation for suspension microlaryngoscopy. J Voice. 2005 Mar;19(1):146-50. doi: 10.1016/j.jvoice.2004.03.008. PMID 15766860
- [Background] Hess MM, Fleischer S, Ernstberger M. New 445 nm blue laser for laryngeal surgery combines photoangiolytic and cutting properties. Eur Arch Otorhinolaryngol. 2018 Jun;275(6):1557-1567. doi: 10.1007/s00405-018-4974-8. Epub 2018 Apr 19. PMID 29675755
- [Background] Helmstaedter V, Tellkamp R, Schwab B, Lenarz T, Durisin M. [High-frequency jet ventilation in otorhinolaryngology - surgical and anaesthesiologic issues]. Laryngorhinootologie. 2014 Jul;93(7):455-60. doi: 10.1055/s-0034-1370925. Epub 2014 Mar 27. German. PMID 24676871
- [Background] Jaquet Y, Monnier P, Van Melle G, Ravussin P, Spahn DR, Chollet-Rivier M. Complications of different ventilation strategies in endoscopic laryngeal surgery: a 10-year review. Anesthesiology. 2006 Jan;104(1):52-9. doi: 10.1097/00000542-200601000-00010. PMID 16394690
- [Background] Heinze H, Eichler W, Karsten J, Sedemund-Adib B, Heringlake M, Meier T. Functional residual capacity-guided alveolar recruitment strategy after endotracheal suctioning in cardiac surgery patients. Crit Care Med. 2011 May;39(5):1042-9. doi: 10.1097/CCM.0b013e31820eb736. PMID 21336125
- [Background] Greene KE, King TE Jr, Kuroki Y, Bucher-Bartelson B, Hunninghake GW, Newman LS, Nagae H, Mason RJ. Serum surfactant proteins-A and -D as biomarkers in idiopathic pulmonary fibrosis. Eur Respir J. 2002 Mar;19(3):439-46. doi: 10.1183/09031936.02.00081102. PMID 11936520
- [Background] Haagsman HP, Hogenkamp A, van Eijk M, Veldhuizen EJ. Surfactant collectins and innate immunity. Neonatology. 2008;93(4):288-94. doi: 10.1159/000121454. Epub 2008 Jun 5. PMID 18525212
- [Background] Wulf-Johansson H, Thinggaard M, Tan Q, Johansson SL, Schlosser A, Christensen K, Holmskov U, Sorensen GL. Circulating surfactant protein D is associated to mortality in elderly women: a twin study. Immunobiology. 2013 May;218(5):712-7. doi: 10.1016/j.imbio.2012.08.272. Epub 2012 Aug 20. PMID 22999473
- [Background] Aihara K, Oga T, Harada Y, Chihara Y, Handa T, Tanizawa K, Watanabe K, Tsuboi T, Hitomi T, Mishima M, Chin K. Comparison of biomarkers of subclinical lung injury in obstructive sleep apnea. Respir Med. 2011 Jun;105(6):939-45. doi: 10.1016/j.rmed.2011.02.016. Epub 2011 Mar 12. PMID 21402472
- [Background] Determann RM, Royakkers AA, Haitsma JJ, Zhang H, Slutsky AS, Ranieri VM, Schultz MJ. Plasma levels of surfactant protein D and KL-6 for evaluation of lung injury in critically ill mechanically ventilated patients. BMC Pulm Med. 2010 Feb 16;10:6. doi: 10.1186/1471-2466-10-6. PMID 20158912
- [Background] Broeckaert F, Clippe A, Knoops B, Hermans C, Bernard A. Clara cell secretory protein (CC16): features as a peripheral lung biomarker. Ann N Y Acad Sci. 2000;923:68-77. doi: 10.1111/j.1749-6632.2000.tb05520.x. PMID 11193780
- [Background] Serpa Neto A, Campos PP, Hemmes SN, Bos LD, Bluth T, Ferner M, Guldner A, Hollmann MW, India I, Kiss T, Laufenberg-Feldmann R, Sprung J, Sulemanji D, Unzueta C, Melo MF, Weingarten TN, Boer AM, Pelosi P, Gama de Abreu M, Schultz MJ; PROVE Network Investigators. Kinetics of plasma biomarkers of inflammation and lung injury in surgical patients with or without postoperative pulmonary complications. Eur J Anaesthesiol. 2017 Apr;34(4):229-238. doi: 10.1097/EJA.0000000000000614. PMID 28187051
- [Background] Hofbauer KH, Jensen BL, Kurtz A, Sandner P. Tissue hypoxygenation activates the adrenomedullin system in vivo. Am J Physiol Regul Integr Comp Physiol. 2000 Feb;278(2):R513-9. doi: 10.1152/ajpregu.2000.278.2.R513. PMID 10666155
- [Background] da Rosa DP, Forgiarini LF, Baronio D, Feijo CA, Martinez D, Marroni NP. Simulating sleep apnea by exposure to intermittent hypoxia induces inflammation in the lung and liver. Mediators Inflamm. 2012;2012:879419. doi: 10.1155/2012/879419. Epub 2012 Nov 26. PMID 23226929
- [Background] Wrigge H, Uhlig U, Baumgarten G, Menzenbach J, Zinserling J, Ernst M, Dromann D, Welz A, Uhlig S, Putensen C. Mechanical ventilation strategies and inflammatory responses to cardiac surgery: a prospective randomized clinical trial. Intensive Care Med. 2005 Oct;31(10):1379-87. doi: 10.1007/s00134-005-2767-1. Epub 2005 Aug 17. PMID 16132888
- [Background] Wrigge H, Uhlig U, Zinserling J, Behrends-Callsen E, Ottersbach G, Fischer M, Uhlig S, Putensen C. The effects of different ventilatory settings on pulmonary and systemic inflammatory responses during major surgery. Anesth Analg. 2004 Mar;98(3):775-81, table of contents. doi: 10.1213/01.ane.0000100663.11852.bf. PMID 14980936
- [Background] Zhang X, Xie M, Gao Y, Wei HH, Zheng JQ. [Study on the effect and mechanism of hypoxia on the histological structure of rat's lung]. Sichuan Da Xue Xue Bao Yi Xue Ban. 2012 Jan;43(1):1-5. Chinese. PMID 22455120